CLINICAL TRIAL: NCT02572167
Title: A Phase 1/2 Study Evaluating Brentuximab Vedotin in Combination With Nivolumab in Patients With Relapsed or Refractory Hodgkin Lymphoma After Failure of Frontline Therapy
Brief Title: A Study of Brentuximab Vedotin Combined With Nivolumab for Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-025
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Hodgkin Lymphoma
Keywords: Monomethyl auristatin E; Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Immunotherapy; Autologous stem cell transplant
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab Vedotin + Nivolumab (Experimental): Brentuximab vedotin plus nivolumab
  Interventions: Drug: brentuximab vedotin; Drug: nivolumab

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg by intravenous (IV) infusion for up to 4 cycles
  Other Names: SGN-35, ADCETRIS
Drug: nivolumab — 3 mg/kg by intravenous (IV) infusion for up to 4 cycles
  Other Names: BMS-936558, OPDIVO

SUMMARY:
The purpose of this study is to assess the safety profile and antitumor activity of brentuximab vedotin administered in combination with nivolumab in patients with relapsed or refractory Hodgkin lymphoma (HL)

DETAILED DESCRIPTION:
This study will examine the safety profile and antitumor activity when brentuximab vedotin is combined with nivolumab. Patients will be treated for up to four 21-day cycles with brentuximab vedotin 1.8 mg/kg and nivolumab 3 mg/kg.

There will be 3 parts to this study. In Part 1, the safety of combination treatment will be evaluated by a Safety Monitoring Committee (SMC) prior to expansion of enrollment to evaluate treatment effect in Part 2. Part 2 of the study will further characterize the safety and antitumor activity of brentuximab vedotin combined with nivolumab by enrolling patients at the recommended dose schedule determined in Part 1. Part 3 of the study will evaluate the safety and antitumor activity of combination treatment administered at an alternate dosing schedule determined by cumulative safety and activity data from Parts 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory Hodgkin lymphoma following failure of standard frontline chemotherapy for the treatment of classical Hodgkin lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Previously treated with brentuximab vedotin, immune-oncology agents, or received an allogeneic or autologous stem cell transplant
* Documented history of a cerebral vascular event
* History of another invasive malignancy that has not been in remission for at least 3 years
* History of progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Galderisi, DO, Study Director — Seagen Inc.
Locations (13):
- United States (13):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - James Cancer Hospital / Ohio State University, Columbus, Ohio
  - Charles A. Sammons Cancer Center / Baylor University Medical Center, Dallas, Texas

REFERENCES:
- [Result] Herrera AF, Moskowitz AJ, Bartlett NL, Vose JM, Ramchandren R, Feldman TA, LaCasce AS, Ansell SM, Moskowitz CH, Fenton K, Ogden CA, Taft D, Zhang Q, Kato K, Campbell M, Advani RH. Interim results of brentuximab vedotin in combination with nivolumab in patients with relapsed or refractory Hodgkin lymphoma. Blood. 2018 Mar 15;131(11):1183-1194. doi: 10.1182/blood-2017-10-811224. Epub 2017 Dec 11. PMID 29229594
- [Derived] Advani RH, Moskowitz AJ, Bartlett NL, Vose JM, Ramchandren R, Feldman TA, LaCasce AS, Christian BA, Ansell SM, Moskowitz CH, Brown L, Zhang C, Taft D, Ansari S, Sacchi M, Ho L, Herrera AF. Brentuximab vedotin in combination with nivolumab in relapsed or refractory Hodgkin lymphoma: 3-year study results. Blood. 2021 Aug 12;138(6):427-438. doi: 10.1182/blood.2020009178. PMID 33827139

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Staggered Dose; Part 2: Staggered Dose Expansion: Brentuximab vedotin plus nivolumab; staggered dose in Cycle 1 only. brentuximab vedotin: 1.8 mg/kg by intravenous (IV) infusion for up to 4 cycles nivolumab: 3 mg/kg by intravenous (IV) infusion for up to 4 cycles
- Part 3: Same-day Dose: Brentuximab vedotin plus nivolumab brentuximab vedotin: 1.8 mg/kg by intravenous (IV) infusion for up to 4 cycles nivolumab: 3 mg/kg by intravenous (IV) infusion for up to 4 cycles
Period: Overall Study
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose
Started | 6 | 56 | 31
Completed | 0 | 0 | 0
Not Completed | 6 | 56 | 31
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Lost to Follow-up | 2 | 5 | 3
Not completed — Death | 0 | 8 | 3
Not completed — Did not meet inclusion criteria | 0 | 0 | 1
Not completed — Study closure by Sponsor | 4 | 40 | 24

BASELINE CHARACTERISTICS:
Population: All Treated Subjects analysis set includes all subjects who received any amount of brentuximab vedotin or nivolumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose | Total
Number analyzed (Participants) | 6 | 55 | 30 | 91
Age, Continuous [Median (Full Range); unit: years] | 26.0 [20 to 37] | 37.0 [18 to 69] | 31.5 [20 to 66] | 34.0 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 27 | 19 | 51
  Male | 1 | 28 | 11 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 9 | 14
  Not Hispanic or Latino | 5 | 49 | 20 | 74
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 6 | 47 | 24 | 77
  More than one race | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 1 | 1 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Measure Description: 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0 | 4 | 35 | 19 | 58
    Grade 1 | 2 | 20 | 10 | 32
    Unknown | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-emergent adverse events (TEAEs) are presented and defined as newly occurring (not present at baseline) or worsening after first dose of investigational product. The timeframe includes a 6.01 month safety reporting period and additional long-term follow up through 28.9 months.
Time Frame: Up to 28.9 months
Population: The safety analysis set includes all patients who receive any amount of brentuximab vedotin or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose
Number analyzed (Participants) | 6 | 55 | 30
Participants
  Any treatment-emergent adverse event (TEAE) | 6 | 55 | 30
  AEs related to brentuximab vedotin only | 5 | 41 | 15
  AEs related to nivolumab only | 3 | 20 | 13
  AEs related to both study drugs | 5 | 37 | 27
  Any serious adverse event (SAE) | 0 | 16 | 5
  SAEs related to brentuximab vedotin only | 0 | 2 | 0
  SAE related to nivolumab only | 0 | 4 | 0
  SAE related to both study drugs | 0 | 5 | 4
  AEs leading to treatment discontinuation | 0 | 1 | 1

2. Primary Outcome: Complete Remission Rate
Description: Number of patients with complete metabolic response (CMR) at end of treatment
Time Frame: Up to 3.42 months
Population: The Efficacy Evaluable analysis set includes all patients who had an adequate baseline disease assessment, received any amount of either drug, and subsequently had an adequate response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose
Number analyzed (Participants) | 6 | 54 | 30
Participants | 4 | 33 | 24

3. Secondary Outcome: Objective Response Rate
Description: Number of patients with complete metabolic response (CMR) or partial metabolic response (PMR)
Time Frame: Up to 3.42 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose
Number analyzed (Participants) | 6 | 54 | 30
Participants | 6 | 43 | 28

4. Secondary Outcome: Duration of Complete Response
Description: The time from start of the first documentation of complete response (CR) to the first documentation of tumor progression (PD) including radiographic evidence of progression and clinical progression per investigator or to death due to any cause, whichever comes first.
Time Frame: Up to 69.3 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose
Number analyzed (Participants) | 4 | 33 | 24
Months | NA [0 to 69.3] — The median duration of CR was not reached for any part of this study. | NA [0 to 61.9] — The median duration of CR was not reached for any part of this study. | NA [0 to 50.4] — The median duration of CR was not reached for any part of this study.

5. Secondary Outcome: Duration of Objective Response
Description: The time from start of the first documentation of OR (CR or PR) to the first documentation of PD or to death due to any cause, whichever comes first.
Time Frame: Up to 69.3 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose
Number analyzed (Participants) | 6 | 43 | 28
Months | NA [0 to 69.3] — The median duration of OR was not reached for any part of this study. | NA [0 to 61.9] — The median duration of OR was not reached for any part of this study. | NA [0 to 50.4] — The median duration of OR was not reached for any part of this study.

6. Secondary Outcome: Progression-free Survival Post-autologous Stem Cell Transplant
Description: For participants who undergo ASCT, the time from ASCT to the first documentation of PD or to death due to any cause, whichever comes first.
Time Frame: Up to 67.3 months
Population: Subset includes all patients who received any amount of brentuximab vedotin or nivolumab and who received a stem cell transplant without intervening salvage after study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-Day Dose
Number analyzed (Participants) | 6 | 36 | 25
Months | NA [0 to 67.3] — The median duration of PFS was not reached for any part of this study. | NA [0 to 61.1] — The median duration of PFS was not reached for any part of this study. | NA [0 to 48.8] — The median duration of PFS was not reached for any part of this study.

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were followed up to 6.01 months. Serious adverse events and all-cause mortality were followed up to 72 months.
Description: All-Cause Mortality includes all patients enrolled in the study.
  Serious Adverse Events and Other Adverse Events includes the safety analysis set - all patients who received any amount of brentuximab vedotin or nivolumab.
Arm/Group | Part 1: Staggered Dose | Part 2: Staggered Dose Expansion | Part 3: Same-day Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 8/56 | 3/31
Serious Adverse Events (participants affected / at risk) | 0/6 | 16/55 | 5/30
Other Adverse Events (participants affected / at risk) | 6/6 | 55/55 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Staggered Dose (N=6) | Part 2: Staggered Dose Expansion (N=55) | Part 3: Same-day Dose (N=30)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Necrotising soft tissue infection (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Systemic candida (Infections and infestations) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 3 | 1
Malaise (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Guillain-barre syndrome (Nervous system disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Staggered Dose (N=6) | Part 2: Staggered Dose Expansion (N=55) | Part 3: Same-day Dose (N=30)
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 30 | 15
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 13 | 11
Rash (Skin and subcutaneous tissue disorders) | 1 | 14 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 12 | 6
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 11 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 9 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 9 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 6 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fatigue (General disorders) | 6 | 39 | 28
Pyrexia (General disorders) | 2 | 24 | 16
Chills (General disorders) | 1 | 16 | 11
Chest discomfort (General disorders) | 0 | 9 | 5
Pain (General disorders) | 0 | 5 | 9
Non-cardiac chest pain (General disorders) | 1 | 4 | 5
Oedema peripheral (General disorders) | 1 | 7 | 1
Asthenia (General disorders) | 0 | 6 | 1
Puncture site pain (General disorders) | 0 | 2 | 3
Malaise (General disorders) | 0 | 2 | 2
Catheter site pain (General disorders) | 0 | 3 | 0
Face oedema (General disorders) | 0 | 1 | 2
Catheter site rash (General disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 41 | 28
Diarrhoea (Gastrointestinal disorders) | 5 | 32 | 22
Vomiting (Gastrointestinal disorders) | 6 | 25 | 18
Constipation (Gastrointestinal disorders) | 3 | 22 | 13
Stomatitis (Gastrointestinal disorders) | 4 | 19 | 12
Abdominal pain (Gastrointestinal disorders) | 1 | 14 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 12 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 9 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 10 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 5 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 4 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 3 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 29 | 20
Anaemia (Blood and lymphatic system disorders) | 6 | 24 | 16
Neutropenia (Blood and lymphatic system disorders) | 6 | 19 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 12 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 7 | 7
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 20 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 15 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 21 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 19 | 10
Dizziness (Nervous system disorders) | 1 | 13 | 4
Paraesthesia (Nervous system disorders) | 1 | 7 | 3
Dysgeusia (Nervous system disorders) | 0 | 4 | 0
Presyncope (Nervous system disorders) | 0 | 4 | 2
Syncope (Nervous system disorders) | 1 | 4 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 4 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 15 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 9 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 11 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 15 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 10 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 8 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 25 | 14
Insomnia (Psychiatric disorders) | 0 | 14 | 10
Depression (Psychiatric disorders) | 1 | 7 | 4
Agitation (Psychiatric disorders) | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 25 | 11
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 2
Hypotension (Vascular disorders) | 2 | 11 | 9
Flushing (Vascular disorders) | 1 | 10 | 3
Hypertension (Vascular disorders) | 0 | 11 | 3
Hot flush (Vascular disorders) | 2 | 5 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 5 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 7 | 5
Nasopharyngitis (Infections and infestations) | 0 | 2 | 3
Folliculitis (Infections and infestations) | 1 | 2 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2
Rash pustular (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 4 | 2
Alanine aminotransferase increased (Investigations) | 0 | 4 | 2
Weight decreased (Investigations) | 0 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2
Weight increased (Investigations) | 0 | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 3
International normalised ratio increased (Investigations) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 9 | 4
Palpitations (Cardiac disorders) | 0 | 3 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 3 | 2
Dysuria (Renal and urinary disorders) | 0 | 5 | 3
Haematuria (Renal and urinary disorders) | 0 | 3 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 2
Polyuria (Renal and urinary disorders) | 0 | 3 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 5 | 2
Engraftment syndrome (Immune system disorders) | 0 | 3 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 4 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2
Thyroiditis (Endocrine disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 4 | 1
Vision blurred (Eye disorders) | 0 | 1 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 4
Thrombosis in device (Product Issues) | 0 | 0 | 2
Swelling face (General disorders) | 0 | 3 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT02572167/Prot_002.pdf
  • Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT02572167/SAP_000.pdf